CLINICAL TRIAL: NCT04813133
Title: Role of Synchronized Lifestyle Modification Program in Peripheral Neuropathy in Insulin Dependent Type 2 Diabetics
Brief Title: Role of Synchronized Lifestyle Modification Program in Insulin Dependent Diabetic Peripheral Neuropathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRC/23/233 Tayyaba Anis Ch.
Record Dates: First submitted 2021-02-02; First posted 2021-03-24 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Neuropathies
Keywords: Synchronized Lifestyle Modification Program; Diabetic Neuropathy; Insulin
MeSH Terms: conditions — Diabetic Neuropathies; Insulin Resistance | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Synchronized Lifestyle Modification Program (Experimental): Synchronized Lifestyle Modification Program
  Interventions: Other: Synchronized Lifestyle Modification Program
- Synchronized Lifestyle Modification Program and Physiotherapy (Experimental): Synchronized Lifestyle Modification Program and Physiotherapy
  Interventions: Other: Synchronized Lifestyle Modification Program and Physiotherapy
- Physiotherapy (Experimental): Physiotherapy included Aerobics, Resistance exercise, Flexibility exercise, and Balance exercise.
  Interventions: Other: Physiotherapy
- Control Group (No Intervention): No intervention will be given to this Group

INTERVENTIONS:
Other: Synchronized Lifestyle Modification Program — Synchronization of dietary intake with circadian rhythm of the body.
  Arms: Synchronized Lifestyle Modification Program
Other: Synchronized Lifestyle Modification Program and Physiotherapy — Synchronization of dietary intake with circadian rhythm of the body along with Physiotherapy ( Aerobics, flexibility, resistance and balance exercises.)
  Arms: Synchronized Lifestyle Modification Program and Physiotherapy
Other: Physiotherapy — Only Physiotherapy training which includes ( Aerobics, flexibility, resistance and balance exercises.)
  Arms: Physiotherapy

SUMMARY:
This study aims to determine the role of Synchronized Lifestyle modification program along with Physiotherapy on the symptoms of DPN in patients on insulin therapy.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a metabolic disorder which influence about 8.3% of adult population and is the fifth major cause of death globally. In Pakistan, prevalence of type 2 diabetes is 16.98% according to recent survey held in 2019. DM is classified into type 1 and type 2 diabetes. In type 1 diabetes, there is an absolute deficiency of insulin secretion due to an autoimmune pathologic process occurring in beta islets of pancreas. While Type 2 diabetes is characterized by a combination of insulin resistance and inadequate insulin secretion with resultant hyperglycemia leading to micro and macrovascular complications. Macrovascular complications include cardiovascular disease, stroke and peripheral artery disease. Amongst microvascular complications, Diabetic peripheral neuropathy (DPN) is one of the most common complication in both developed and developing countries. DPN is a symmetrical, length-dependent sensorimotor polyneuropathy which is attributed to metabolic and micro vessel alterations due to hyperglycemia and concomitant cardiovascular risk covariates. Major risk factors for development of DPN include duration of diabetes, hyperglycemia, and age, followed by prediabetes, hypertension, dyslipidemia, and obesity. DPN can engender disablement in touch sensation, vibration sense, lower limb proprioception, and kinesthesia thus contributing to impaired balance, altered gait with increased risk of falling. DPN occurs in more than 50% of people with type 2 diabetes. It is a salient risk factor for skin breakdown, amputation, and reduced physical mobility consequently lowering the quality of life Management of DPN is multifaceted and includes efforts to alter the natural history (lifestyle changes) and symptomatic treatments through pharmacological interventions. Daily habits and actions exert an enormous influence on short-term and long-term health and quality of life. Importance of dietary modification is enhanced if it is synchronized with the circadian rhythm of the body. Therefore, Synchronized Lifestyle modification program is a personalized, homeostasis restoring, liver centric lifestyle modification program that works through the correction of body clock rhythm. Lifestyle medicine comprises of cluster of positive lifestyle practices including maintenance of a healthy body weight, regular physical activity, cessation of cigarette smoking, stress reduction as well following a few nutritional practices such as increasing whole grains and consuming more fruits and vegetables. Lifestyle modification, including diet and exercise, slow the progression of neuropathy by promoting small nerve fiber regeneration. Dietary modifications include intake of nutrient, such as whole grains, vegetables, fruits, legumes, low-fat dairy, lean meats, nuts, and seeds. These foods help to maintain body weight, attain individualized glycemic, blood pressure, and lipid goals and prevent complications of diabetes. Exercise improves three of the biggest risk factors for diabetic neuropathy including insulin sensitivity and glucose control, obesity, and dyslipidemia. These exercises include aerobic exercise that improves glycemic control and insulin sensitivity in diabetics. Strength training exercise improves postural sway during standing, and gait characteristics during level-ground walking. While the flexibility exercise are suggested for refining distal joint mobility and plantar pressure distribution during gait. Thus, Exercise is known to enhance multiple metabolic factors that may affect nerve health and microvascular function, which may indirectly protect against peripheral nerve damage.

ELIGIBILITY:
Inclusion Criteria:

1. Both males and females
2. Five years duration of clinically diagnosed type 2 Diabetes were included in the study
3. On insulin therapy
4. Diagnosed to have peripheral neuropathy according to Michigan Neuropathy Screening Instrument with a physical examination score > 2.5

Exclusion Criteria:

1. Type 1 Diabetics
2. Type 2 Diabetics
3. On oral hypoglycemic and Glucagon-like Peptide-1 analogues, patients having neuropathies due to other causes (Vitamin B₁₂ deficiency, Drug and Alcohol abuse), patients with other co-morbidities (Renal insufficiency, Heart, Liver and Eye diseases)
4. Patients with foot ulcers and orthopedic or surgical problems of lower limb
5. Patients with peripheral vascular diseases, inability to walk independently
6. Patients receiving any structured supervised physiotherapy intervention
7. Pregnant females were excluded from the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Lifestyle pattern assessment | 12 weeks
  Changes from baseline assessed through a self structured questionnaire consisted of open ended questions to assess the timing and type of food taken in meals, daily water intake and sleeping habits. Total 10 questions are included.
Calculation of Body Mass Index | 12 weeks
  Changes from baseline calculated by measuring height through metal measuring tape in meters and weight in kilograms through potable manual weighing scale. BMI with minimum value of 18.5 and maximum value of 24.5 Kilogram/ square meter. Below 18.5 is considered as underweight and above 24.9 is considered as obese
Measurement of Systolic Blood Pressure | 12 weeks
  Changes from baseline are assessed by using Mercury Sphygmomanometer with minimum value of 110 millimeter of Mercury and maximum value of 130 millimeter of Mercury. Below 110 millimeter of Mercury is considered as low systolic pressure and above 130 millimeter of Mercury is considered as high systolic pressure
Measurement of Diastolic Blood Pressure | 12 weeks
  Changes from baseline are assessed by using Mercury Sphygmomanometer with minimum value of 60 millimeter of Mercury and maximum value of 90 millimeter of Mercury. Below 60 millimeter of Mercury is considered as low diastolic pressure and above 90 millimeter of Mercury is considered as high diastolic pressure
Assessment of Presence and Severity of Neuropathy by Michigan Neuropathy Screening Instrument (MNSI) | 12 weeks
  Changes from baseline are assessed by Michigan Neuropathy Screening Instrument (MNSI) that consists of a history questionnaire comprising of 15 questions related to symptoms of diabetic neuropathy with a score of >7 is considered as abnormal and Physical examination that consists of inspection of foot for deformities, ulcers and callus formation, Ankle reflex and vibration sensation with a score of >2.5 is considered abnormal
Measurement of Peak Latency of Sensory Nerves of lower extremities (Sural and Peroneal) | 12 weeks
  Changes from baseline are assessed by Nerve Conduction Studies with a maximum value of 4.2 millisecond for sural nerve and 6.1 milliseconds for peroneal nerve are considered normal. Values below 4.2 and 6.1 milliseconds are considered abnormal.
Measurement of Amplitude of Sensory Nerves of lower extremities (Sural and Peroneal) | 12 weeks
  Changes from baseline are assessed by Nerve Conduction Studies with a value of 2 microvolts for peroneal nerve and 6 microvolts for sural nerve are considered normal. Values below 2 and 6 microvolts were considered abnormal.
Velocity of Sensory Nerves of lower extremities (Sural and Peroneal) | 12 weeks
  Changes from baseline are assessed by Nerve Conduction Studies with minimum limit of 44 meters /second and maximum limit of 64 meters/second. Value below 44m/sec and above 64m/sec are considered abnormal.
Onset Latency of Motor Nerves (Peroneal and Tibial) | 12 weeks
  Changes from baseline are assessed by Nerve Conduction Studies with a value of 6.1 milliseconds for both nerves is considered normal. Value below 6.1 milliseconds is considered abnormal.
Amplitude of Motor Nerves (Peroneal and Tibial) | 12 weeks
  Changes from baseline are assessed by Nerve Conduction Studies with a value of 2 millivolts for peroneal nerve and 3 millivolts for tibial nerve is considered normal. Value below 2 and 3 microvolts is considered abnormal.
Velocity of Motor Nerves (Peroneal and Tibial) | 12 weeks
  Changes from baseline are assessed by Nerve Conduction Studies with a value of 41 m/sec is considered normal. Value below 41 m/sec is considered abnormal
Assessment of Balance by Berg Balance Scale (BBS) | 12 weeks
  Changes from baseline are assessed by Berg Balance Scale (BBS) with Low Fall Risk score of 41-56, Medium Fall Risk 21-40, High Fall Risk 0-20
Fasting Blood Glucose | 12 weeks
  Changes from baseline are measured by glucose oxidase strip method in milligram/deciliter using glucometer with a minimum value of 72 mg/dL and a maximum value of 99mg/dL is considered normal. Value below 72mg/dL is considered as hypoglycemia and value above 99 mg/dL is considered hyperglycemia.
Serum HbA1c concentration | 12 weeks
  Changes from baseline are measured by Ion Exchange Chromatography with a minimum value of 4% and maximum value of 5.9% is considered normal.
Serum Triglycerides | 12 week
  Changes from baseline are measured by Glycerol Phosphate Enzyme Based Method with a minimum value of 150 milligram /deciliter and a maximum value of 199 milligram/deciliter is considered normal. Value above 200 milligram/deciliter is considered as increased serum triglycerides
Serum Total Cholesterol | 12 weeks
  Changes from baseline are measured by Cholesterol Oxidase Enzyme Based Method with a minimum value of 125 and a maximum value of 200 milligram /deciliters considered as normal. Value above 200 milligram/deciliter is considered as hypercholesterolemia.
Serum Low Density Lipoproteins (LDL) | 12 weeks
  Changes from baseline are measured by Friedewald calculation with a minimum value of 100 and a maximum value of 120 milligram /deciliter is considered as normal.
Serum High Density Lipoproteins (HDL) | 2 weeks
  Changes from baseline are measured by Direct Enzymatic Immuno-inhibition with a maximum value of 40milligram/deciliter and higher is considered as normal. Value below 40 milligram/deciliter is considered as abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Shazia Ali, PhD, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway Hospital, Islamabad, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Domingueti CP, Dusse LM, Carvalho Md, de Sousa LP, Gomes KB, Fernandes AP. Diabetes mellitus: The linkage between oxidative stress, inflammation, hypercoagulability and vascular complications. J Diabetes Complications. 2016 May-Jun;30(4):738-45. doi: 10.1016/j.jdiacomp.2015.12.018. Epub 2015 Dec 18. PMID 26781070
- [Background] Aamir AH, Ul-Haq Z, Mahar SA, Qureshi FM, Ahmad I, Jawa A, Sheikh A, Raza A, Fazid S, Jadoon Z, Ishtiaq O, Safdar N, Afridi H, Heald AH. Diabetes Prevalence Survey of Pakistan (DPS-PAK): prevalence of type 2 diabetes mellitus and prediabetes using HbA1c: a population-based survey from Pakistan. BMJ Open. 2019 Feb 21;9(2):e025300. doi: 10.1136/bmjopen-2018-025300. PMID 30796126
- [Background] Diabetes DOF. DEFINITION AND DESCRIPTION OF DIABETES OTHER CATEGORIES OF GLUCOSE. 2010;33.
- [Background] Lilly E, Homburg B. P R O G R E S S I O N , Initiating Insulin Therapy in Type 2. 2009;32:0-5.
- [Background] Majeedkutty NA, Jabbar MA. Physical Therapy for Diabetic Peripheral Neuropathy : A Narrative Review. 30(1):112-25.
- [Background] Alam U, Riley DR, Jugdey RS, Azmi S, Rajbhandari S, D'Aout K, Malik RA. Diabetic Neuropathy and Gait: A Review. Diabetes Ther. 2017 Dec;8(6):1253-1264. doi: 10.1007/s13300-017-0295-y. Epub 2017 Sep 1. PMID 28864841
- [Background] Papanas N, Ziegler D. Risk Factors and Comorbidities in Diabetic Neuropathy: An Update 2015. Rev Diabet Stud. 2015 Spring-Summer;12(1-2):48-62. doi: 10.1900/RDS.2015.12.48. Epub 2015 Aug 10. PMID 26676661
- [Background] Kluding PM, Bareiss SK, Hastings M, Marcus RL, Sinacore DR, Mueller MJ. Physical Training and Activity in People With Diabetic Peripheral Neuropathy: Paradigm Shift. Phys Ther. 2017 Jan 1;97(1):31-43. doi: 10.2522/ptj.20160124. PMID 27445060
- [Background] Education DS. 4 . Lifestyle Management. 2017;40(January):33-43.
- [Background] Nadi M, Marandi SM, Esfarjani F, Saleki M, Mohammadi M. The Comparison between Effects of 12 weeks Combined Training and Vitamin D Supplement on Improvement of Sensory-motor Neuropathy in type 2 Diabetic Women. Adv Biomed Res. 2017 May 2;6:55. doi: 10.4103/2277-9175.205528. eCollection 2017. PMID 28553628
- [Background] Handsaker JC, Brown SJ, Bowling FL, Maganaris CN, Boulton AJ, Reeves ND. Resistance exercise training increases lower limb speed of strength generation during stair ascent and descent in people with diabetic peripheral neuropathy. Diabet Med. 2016 Jan;33(1):97-104. doi: 10.1111/dme.12841. Epub 2015 Jul 17. PMID 26108438
- [Background] Andayani TM, Izham M, Ibrahim M, Asdie AH. Comparison of the glycemic control of insulin and triple oral therapy in type 2 diabetes mellitus. 2010;1(April):13-8.
- [Background] Rahimi N, Samavati Sharif MA, Goharian AR, Pour AH. The Effects of Aerobic Exercises and 25(OH) D Supplementation on GLP1 and DPP4 Level in Type II Diabetic Patients. Int J Prev Med. 2017 Aug 8;8:56. doi: 10.4103/ijpvm.IJPVM_161_17. eCollection 2017. PMID 28900535
- [Background] DE BODO RC, ALTSZULER N, DUNN A, STEELE R, ARMSTRONG DT, BISHOP JS. Effects of exogenous and endogenous insulin on glucose utilization and production. Ann N Y Acad Sci. 1959 Sep 25;82:431-51. doi: 10.1111/j.1749-6632.1959.tb44924.x. No abstract available. PMID 13814676
- [Background] Donnor T, Sarkar S. Insulin- Pharmacology, Therapeutic Regimens and Principles of Intensive Insulin Therapy. 2023 Feb 15. In: Feingold KR, Adler RA, Ahmed SF, Anawalt B, Blackman MR, Chrousos G, Corpas E, de Herder WW, Dhatariya K, Dungan K, Hamilton E, Hofland J, Jan de Beur S, Kalra S, Kaltsas G, Kapoor N, Kim M, Koch C, Kopp P, Korbonits M, Kovacs CS, Kuohung W, Laferrere B, Levy M, McGee EA, McLachlan R, Muzumdar R, Purnell J, Rey R, Sahay R, Shah AS, Sperling MA, Stratakis CA, Trence DL, Wilson DP, editors. Endotext [Internet]. South Dartmouth (MA): MDText.com, Inc.; 2000-. Available from http://www.ncbi.nlm.nih.gov/books/NBK278938/ PMID 25905175